CLINICAL TRIAL: NCT07210151
Title: Anatomical Navigation for Guided Electrophysiology in AFL and AFib
Acronym: ANGEL-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LUMA Vision Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANGEL-AF -P004
Record Dates: First submitted 2025-09-19; First posted 2025-10-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Atrial Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atrial Fibrillation and Atrial Flutter arm (Experimental): Subjects entitled to undergo a catheter-based ablation treatment for typical atrial flutter and/or atrial fibrillation
  Interventions: Device: VERAFEYE Anatomic Guidance System

INTERVENTIONS:
Device: VERAFEYE Anatomic Guidance System — The VERAFEYE Anatomical Guidance System will be used during standard of care, catheter-based treatments for atrial flutter and/or atrial fibrillation.

SUMMARY:
The objective of the study is to collect data on the use of the VERAFEYE Anatomical Guidance System in adult patients indicated to undergo a catheter ablation procedure for the treatment of Atrial Flutter (AFL), paroxysmal AF (PAF) or persistent AF (perAF).

The study will collect specific information on management of AFL/AF ablation procedures with the commercial VERAFEYE Anatomical Guidance System including but not limited to acute procedural success , and how the VERAFEYE Anatomical Guidance System is used overall. Results from this study may be used to guide development and refinement the VERAFEYE Anatomical Guidance System.

ELIGIBILITY:
Inclusion Criteria:

* IC1: Subject is at least 18 years of age at the time of consent
* IC2: Subject is scheduled to undergo a catheter-ablation procedure to treat AFL/AF (*according to current international and local guidelines and per physician discretion)
* IC3: Subject is able to understand and willing to provide written informed consent
* IC4: Subject is able and willing to complete all study assessments associated with this clinical study at an approved clinical study site

Exclusion Criteria:

* EC1: Subject where placement of VERAFEYE Imaging Catheter is technically not feasible per physician discretion
* EC2: Pregnant women or women who plan to become pregnant during the course of their participation in the study (women should either be of non- childbearing potential at the time of enrolment (as documented in the medical file) or have a negative pregnancy test within the previous 7 days prior to the procedure)
* EC3: Unrecovered/unresolved Adverse Events from any previous invasive procedure
* EC4: Any planned surgical or endovascular intervention within 30 days before or after the ablation procedure.
* EC5: Life expectancy less than 12 months
* EC6: Current LA thrombus

Note: Screening for LA thrombus is required to be performed within 48 hours prior to or during the index procedure. Method of screening per physician discretion. If an atrial thrombus is observed prior to or during the planned index procedure, the index procedure will not begin or will be terminated before accessing the left atrium, and no ablation will be performed. The index procedure for this subject may be rescheduled to be performed within 30 days post ICF signature, provided that the thrombus is no longer present.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Acute procedural success rates during the index procedure | During the procedure
  A procedure will be defined as successful if all the following conditions occur during the case:
  * Ability to create a 3D anatomical model of RA and/or LA with the VERAFEYE Imaging and Guidance System and
  * Ability to complete all necessary ablation lesion sets using the 3D anatomical model of RA and/or LA created with the VERAFEYE System

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce Hospital, Prague, Czechia